CLINICAL TRIAL: NCT01293071
Title: The SATURN Consortium, "Impact of Specific Antibiotic Therapies on the Prevalence of hUman Host ResistaNt Bacteria". Workpackage 2: The SATURN ICU-trial.
Brief Title: Effect of Antibiotic Rotation in the ICU on the Prevalence of Antibiotic Resistant Gram-negative Colonisation
Acronym: SATURN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, MJM Bonten, Prof.dr., UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UMCU_SATURNWP2; 2011-000405-42 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Infections
Keywords: Antibiotic rotation; Cycling; Mixing; Gram-negative; EU; Multi center; Multi Centre; Cluster randomized trial; Cross over
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mixing arm (Active Comparator): Antibiotic rotation, each consecutive initiated antibiotic treatment a different class (one of 3 classes: cephalosporins, piperacillin-tazobactam, carbapenems)
  Interventions: Other: Antibiotic rotation
- Cycling (Active Comparator): Antibiotic rotation, every 1.5 month a different preferred antibiotic treatment from a different class (one of 3 classes: cephalosporins, piperacillin-tazobactam, carbapenems) is used for empiric treatment.
  Interventions: Other: Antibiotic rotation

INTERVENTIONS:
Other: Antibiotic rotation — Rotation of antibiotic classes as specific preferred antibiotic class to be used for empiric treatment of ICU acquired infections.
  Other Names: Any antibiotic from the local guidelines can be used.

SUMMARY:
The SATURN ICU-trial studies the effect of antibiotic rotation on the prevalence of antibiotic resistant Gram-negative colonisation.

DETAILED DESCRIPTION:
Antibiotic rotation has been previously studied with varied results. The theory behind antibiotic rotation is that intermittently changing antibiotic classes will reduce the ecological selective pressure that drives the emergence of antibiotic resistance.

This study compares the effect of 2 types of antibiotic rotation on Gram-negative colonisation in the ICU and also compares both interventions with standard care.

The two interventions apply to the empiric treatment and are: 1) "fast" rotation, i.e. every other patient another class and 2) "slow" rotation, i.e. every other 1.5month another preferred class for empiric Gram-negative antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* There are at least 8 beds, with an average bed-occupancy of 80%; all of which have capacity for mechanical ventilation.
* The ICU can adhere to the selected antibiotics for empiric treatment of infections.
* There is an operational digital patient-information system, from which data can be extracted and delivered in a pre-defined format. Specifically an automated process for digital data-collection regarding microbiological culture-results (from swabs and bacteraemias), antibiotic prescription and patient demographics and illness severity-scores.
* Colonization with ESBL or resistance for any of the antibiotic groups is endemic, with proportions of ICU-acquired bacteraemias used as a proxy. Therefore, the investigators prefer proportions of AMRB infection in the period 2008-2009 to be: ESBL resistance among GNB 1 to 10% Piperacillin/Tazobactam among GNB 1 to10% Carbapenem resistance among Klebsiella Pneumoniae less than 5%
* Have the ability of at least one dedicated Infection Control HCW available for 0,2fte, for patient monitoring, compliance monitoring and instruction of HCWs regarding interventions. In the following this person will be called "Research-Nurse" or "RN".
* Can store screening-cultures at -70ºC
* Can facilitate transport through a UMCU courier.
* There is written approval for the study from the institution's IRB with a waiver for patient informed consent.
* A signature page is signed by the daily management of the candidate-ICU by both ICU physician and director and the ICU nursing-director and presented to the UMCU, indicating willingness to enroll the candidate-ICU in the study.

Exclusion Criteria:

ICUs planning to introduce, during the SATURN trial period, any major diagnostic- or intervention program that will affect AMRB ecology*

* Burn units; due to the specific nature of the care provided and the patients admitted.
* Cardiothoracic surgery units; because of the expected small number of patients admitted for three days or more.
* Paediatric and neonatal ICUs.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean prevalence of ICU patients colonised with antimicrobial resistant Gram-negative pathogens | Monthly point-prevalence screening of all ICU patients

SECONDARY OUTCOMES:
AMRB acquisition incidence, measured as status conversion from noncolonized to colonized during admission at ICU per 100 patients. | 2011-2013
ICU-acquired bacteraemia rate with AMRB (expressed as the rate of ICU-acquired bacteraemia per 1000 patient-days) | 2011-2013
Overall length of ICU-stay hospital-stay and percentage of in-hospital mortality of the total admitted ICU-population. | 2011-2013
Effectiveness of empirical treatment of ICU-acquired bacteraemia, expressed as proportion of bacteraemia for which appropriate antibiotics are administered within 24 hours with antibiotics that the specific pathogens is susceptible for. | 2011-2013

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, MD PhD Professor, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] van Duijn PJ, Verbrugghe W, Jorens PG, Spohr F, Schedler D, Deja M, Rothbart A, Annane D, Lawrence C, Jereb M, Seme K, Sifrer F, Tomic V, Estevez F, Carneiro J, Harbarth S, Bonten MJM. The effects of antibiotic cycling and mixing on acquisition of antibiotic resistant bacteria in the ICU: A post-hoc individual patient analysis of a prospective cluster-randomized crossover study. PLoS One. 2022 May 3;17(5):e0265720. doi: 10.1371/journal.pone.0265720. eCollection 2022. PMID 35503768
- [Derived] van Duijn PJ, Verbrugghe W, Jorens PG, Spohr F, Schedler D, Deja M, Rothbart A, Annane D, Lawrence C, Nguyen Van JC, Misset B, Jereb M, Seme K, Sifrer F, Tomic V, Estevez F, Carneiro J, Harbarth S, Eijkemans MJC, Bonten M; SATURN consortium. The effects of antibiotic cycling and mixing on antibiotic resistance in intensive care units: a cluster-randomised crossover trial. Lancet Infect Dis. 2018 Apr;18(4):401-409. doi: 10.1016/S1473-3099(18)30056-2. Epub 2018 Jan 26. PMID 29396000
- [Derived] van Duijn PJ, Bonten MJ. Antibiotic rotation strategies to reduce antimicrobial resistance in Gram-negative bacteria in European intensive care units: study protocol for a cluster-randomized crossover controlled trial. Trials. 2014 Jul 10;15:277. doi: 10.1186/1745-6215-15-277. PMID 25011604